CLINICAL TRIAL: NCT02952287
Title: Assessment of Flow With the New Four-dimensional Velocity-encoded Magnetic Resonance Imaging Technique
Acronym: 4D Flow
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistically recruitment was not applicable after trial of a few patients
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Shi-Joon Yoo, Cardiac Radiologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REB1000050375
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Congenital Heart Disease (CHD)
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Participants (Experimental): 4D PC MRI acquisition
  Interventions: Device: 4D PC MRI acquisition

INTERVENTIONS:
Device: 4D PC MRI acquisition — Flow-sensitive 4D-MRI acquisitions will be synchronized to the heart rate and breathing using prospective ECG-gating and adaptive diaphragm navigator gating41. The MRI sequence will consist of a segmented k-space spoiled gradient echo sequence with interleaved 3D velocity encoding. Data will be acquired in a sagittal oblique 3D data volume individually adapted to include the heart and the thoracic and upper abdominal vessels of interest like ascending, transverse and descending aorta, main and branch pulmonary arteries, pulmonary veins, superior and inferior vena cava, celiac and superior mesenteric vessels. Velocity encoding (VENC) will be set at 150-500 cm/sec to encompass flow in various vessels.

SUMMARY:
The purpose of our study is to validate the accuracy of 4D PC flow method in quantification of thoracic and upper abdominal blood flow volumes in children. In this validation study, 4D PC flow method will be applied in 100 pediatric patients undergoing clinically indicated CMR with 2D PC flow measurement.

DETAILED DESCRIPTION:
Measurement of blood flow in vessels leading to or arising from the heart is one of the key features of Cardiac Magnetic Resonance (CMR). With standard 2D phase contrast (PC) flow measurements, each vessel is measured separately at a predefined location. Planning and scanning can be time consuming while the patient is inside the scanner. In addition, when the scan time is long, the hemodynamics may be assessed at different physiological states. In contrast to a 2D PC acquisition 4D PC captures all the information about blood flow velocities within a 3D anatomical volume. Once this predefined volume has been acquired, the flow within the heart and vessels of interest can be measured at any desired location offline, i.e. after the patient has left the scanner. This is especially advantageous in cases where multiple 2D PC MRI scans are needed such as in congenital heart disease (CHD). In addition to standard measurements, 4D PC provides flow patterns, which might change our current understanding of pathologic flow conditions. Although there has been increasing interest in this new technique, only a few papers have proved its accuracy in adult population. The purpose of our study is to validate the accuracy of 4D PC flow method in quantification of thoracic and upper abdominal blood flow volumes in children. In this validation study, 4D PC flow method will be applied in 100 pediatric patients undergoing clinically indicated CMR with 2D PC flow measurement.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients under 18 years of age undergoing CMR with 2D PC flow measurements as a clinically indicated component of the examination at The Hospital for Sick Children, Toronto, ON.
* Ability to undergo an MRI examination without anesthesia or sedation.
* Ability to undergo an MRI examination using 'Feed-and-Sleep' technique39

Exclusion Criteria:

* Refusal of consent / assent by parent / legal guardian / patient
* General contraindications for an MRI examination such as non-MRI compatible metallic implants, claustrophobia.
* Patients who require anaesthesia or sedation for MRI

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Pearson´s correlation coefficient (r) | Six months
  The association of variables (stroke volumes as measured with 2D and 4D flow, regurgitation fractions) will be investigated with Pearson´s correlation coefficient (r). P values of <0.05 will be considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Joon Yoo, MD, Principal Investigator — The Hospital for Sick Children

IPD SHARING:
Plan to Share IPD: No